CLINICAL TRIAL: NCT05620238
Title: A Prospective Clinical, Mixed-method Study Exploring Patient and Health Care Perspectives
Brief Title: Home Treatment With Carfilzomib in Patients With Multiple Myeloma
Status: Recruiting | Type: Observational
Sponsor: Thomas Lund (Other)
Responsible Party: Sponsor-Investigator, Thomas Lund, Principal Investigator, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: Home Carfi
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Carfilzomib — Investigate the home administration of Carfilzomib IV reported by both patients and health care staff compared to the hospital setting.
  Other Names: Kyprolis

SUMMARY:
New treatment regimens with increased efficiency and reduced toxicities are being introduced in the treatment of Multiple Myeloma (MM). As a result, patients can expect increased survival, but also increased time on active treatment. Consequently, patients spend an increasing amount of time at the hospital and on transportation. This may not only expose the patients to unnecessary risks of infections, but will also reduce their available time to have a meaningful life. Carfilzomib is a drug used alone or in combination with other drugs for treatment of relapsed multiple myeloma. It is gives as an intravenous infusion day 1 and 2, day 8 and 9, and day 15 and 16 every 28th day. Thus, the patients have to show up at the hospital many times with the risk of acquiring infections. Likewise they sometimes live a long way from the hospital, and therefore spent a lot of time on transportation to and from treatment.

The investigator wish to minimize the number of times the patients have to go to the hospital, by educating them to self-administer day 2, 9 and 16 in their own home. The investigator hope thereby to reduce their risk of hospital-acquired infections and to reduce the time spent on transportation to and from treatment. From a hospital point of view the investigator hope it will reduce the pressure on space in the outpatient clinic; that it will reduce the time a nurse spent on treatment.

In the present project, intravenous Carfilzomib is administered in the hospital through a peripheral intravenous needle on day 1, 8, and 15 of a 28-day cycle and the treatment for the day after is handed to the patient in a cooling compartment. The next day the patient will load the Carfilzomib into the pump and attach it to the peripheral intravenous needle. Once the infusion if finished, the patient will remove the needle and the following week, bring the cooling compartment and the pump back to the hospital.

DETAILED DESCRIPTION:
New treatment regimens with increased efficiency and reduced toxicities are being introduced in the treatment of Multiple Myeloma (MM). As a result, patients can expect increased survival, but also increased time on active treatment. Consequently, patients spend an increasing amount of time at the hospital and on transportation. This may not only expose the patients to unnecessary risks of infections, but will also reduce their available time to have a meaningful life. Carfilzomib is a drug used alone or in combination with other drugs for treatment of relapsed multiple myeloma. It is gives as an intravenous infusion day 1 and 2, day 8 and 9, and day 15 and 16 every 28th day. Thus, the patients have to show up at the hospital many times with the risk of acquiring infections. Likewise they sometimes live a long way from the hospital, and therefore spent a lot of time on transportation to and from treatment.

The investigator wish to minimize the number of times the patients have to go to the hospital, by educating them to self-administer day 2, 9 and 16 in their own home. The investigator hope thereby to reduce their risk of hospital-acquired infections and to reduce the time spent on transportation to and from treatment. From a hospital point of view the investigator hope it will reduce the pressure on space in the outpatient clinic; that it will reduce the time a nurse spent on treatment.

In the present project, intravenous Carfilzomib is administered in the hospital through a peripheral intravenous needle on day 1, 8, and 15 of a 28-day cycle and the treatment for the day after is handed to the patient in a cooling compartment. The next day the patient will load the Carfilzomib into the pump and attach it to the peripheral intravenous needle. Once the infusion if finished, the patient will remove the needle and the following week, bring the cooling compartment and the pump back to the hospital.

Data concerning number of hospital visits, time spend on medication administration, and transportation time will be collected from all 12 patients during cycle 3-4. The investigator will also registered if the patients starts home treatment during cycle 2. In addition, to further explore the patients and the health care professionals' experiences with home treatment, a semi-structured interviews with the first five patients and possibly their relatives, will be conducted once they have received at least 4 cycles. In addition, one focus group interview of the healthcare professionals involved will be conducted once the project have included and treated all 12 patients.

Quantitative data will be presented as counts and percentages for categorical data and as mean and standard deviation or median and interquartile for continuous data. The qualitative data will be analyzed via the method of condensation, in which the essence of the meanings of the interviewees' statements is summarized and subdivided into themes and thereafter into descriptive statements, so that the data is systematically reviewed and divided, and is then able to form the basis for analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Multiple Myeloma in treatment with Carfilzomib
* Patients must have received a minimum of one treatment cycle in the outpatient clinic
* Patients must understand and speak Danish

Exclusion Criteria:

* Patients receiving trial medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Multople Myeloma in treatment with IV Carfilzomib
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Patients satisfaction | 15.12.2022-01.04.2024
  Patients satisfaction reported by semi-structured interviews and Pro-data regarding prefered treatment method

SECONDARY OUTCOMES:
Examination of patients and health care staffs time spent on treatment | 15.12.2022-01.04.2024
  Examination of patients and health care staffs time spent on treatment in minutes on paper

CONTACTS AND LOCATIONS:
Overall Officials: Nana Hyldig, PhD, RN, Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No